CLINICAL TRIAL: NCT06381232
Title: Collection and Analyses of Physiological, Physical, and Molecular Data From a Diverse Population
Status: Recruiting | Type: Observational
Sponsor: Viome (Industry)
Responsible Party: Sponsor
Other Study IDs: VIOME-001
Record Dates: First submitted 2024-04-18; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-03

CONDITIONS: General Health; Wellness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Control
  Interventions: Other: No Intervention
- Cases (Various Phenotypes)
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is an observational study, there are no interventions.

SUMMARY:
The purpose of the study is to collect and analyze physiological, physical, and molecular data from a diverse population to increase our understanding of how such parameters are associated with health and disease.

DETAILED DESCRIPTION:
The analyses conducted by Viome will include, but are not limited to: genetic, transcriptomic, metabolomic, physiological, and physical. The samples collected from participants may include any of these: stool, blood, saliva, cheek swab, vaginal, breast milk/colostrum, nasal swabs or washes, and urine.

Study participants will collect the clinical samples and ship them to Viome labs or CROs (Contract Research Organizations), where they will be analyzed.

The objective of the study is to establish which foods correspond with increased wellness, and which foods correspond to decreased wellness.

The study hypothesis is that by monitoring the patterns of food intake and lifestyle parameters, in conjunction with non-invasive sample testing, personalized diet and lifestyle recommendations can be elucidated.

ELIGIBILITY:
Inclusion Criteria:

* Anyone that resides in the US at the time of enrollment.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants with specific phenotypes of interest and matched healthy controls.
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2018-07-23 (Actual); Primary Completion 2028-07-23 (Estimated); Study Completion 2028-07-23 (Estimated)

PRIMARY OUTCOMES:
Molecular Determinants of Health and Disease | 10 years
  We measure thousands of transcript levels in multiple clinical samples. The primary outcome measures are changes in quantitative gene expression, microbial or human, as a result of transitioning from a healthy state to a disease.

CONTACTS AND LOCATIONS:
Overall Officials: Momchilo Vuyisich, PhD, Principal Investigator — Viome
Locations (1):
- Viome Life Sciences, Bothell, Washington, United States